CLINICAL TRIAL: NCT00828646
Title: Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-708163 in Healthy Male Japanese Subjects and a Comparison to Healthy Elderly Japanese Subjects
Brief Title: Safety Study of Multiple-dose of Gamma-secretase Inhibitor in Healthy Male Japanese and Healthy Elderly Japanese
Acronym: JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN156-012
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-708163 - Panel 1 (Experimental): (Age 20-45 years)
  Interventions: Drug: BMS-708163; Drug: Placebo
- BMS-708163 - Panel 2 (Experimental): (Age 20-45 years)
  Interventions: Drug: BMS-708163; Drug: Placebo
- BMS-708163 - Panel 3 (Experimental): (age 65 or above)
  Interventions: Drug: BMS-708163; Drug: Placebo
- BMS-708163 - Panel 4 (Experimental): (age 65 or above)
  Interventions: Drug: BMS-708163; Drug: Placebo

INTERVENTIONS:
Drug: BMS-708163 — Capsules, Oral, 50 mg, once daily, 14 days
  Arms: BMS-708163 - Panel 1; BMS-708163 - Panel 3
Drug: BMS-708163 — Capsules, Oral, 100 mg/day, once daily, 14 days
  Arms: BMS-708163 - Panel 2
Drug: BMS-708163 — Capsules, Oral, 75 or 100 mg/day, once daily, 14 days
  Arms: BMS-708163 - Panel 4
Drug: Placebo — Capsules, Oral, once daily, 14 days

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, pharmacokinetics, and pharmacodynamics following 14-day multiple oral doses BMS-708163 in healthy young male Japanese and healthy elderly male and female Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 19 to 25 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2
* Men, ages 20 to 45, and men and women [not of childbearing potential (i.e., who are postmenopausal or surgically sterile)], ages 65 or older. Women are considered surgically sterile only if they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy. Women are considered postmenopausal only if they have had amenorrhea for ≥12 consecutive months, or for women on hormone replacement therapy (HRT), if they have a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL

Exclusion Criteria:

* WOCBP
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to administration of investigational product
* Sexually active fertile men not using effective birth control if their partners are WOCBP
* Any significant acute or chronic medical illness
* Any current or recent? medical history of gastrointestinal disease that may affect evaluation of study treatment
* History of recent major surgery or gastrointestinal surgery that may impact on evaluation or absorption of study drug
* History of blood donation or blood transfusion within 4 weeks prior to the study treatment
* Intolerance to oral medication or venous access
* QTc interval (Bazett's correction) >500 ms at screening
* Smoking more than 10 cigarettes per day
* Recent (within 6 months) drug or alcohol abuse as defined in DSM IV
* Any other sound medical, psychiatric and/or social reason as determined by the investigator
* Subjects ≥ 65 yr are allowed to have age-related minimum or mild abnormalities in vital sign (i.e. blood pressure) or laboratory tests (i.e. blood sugar, serum cholesterol, or serum triglyceride) as far as they are not deemed signs or consequences of illness or organ dysfunction and a subject of medical treatment
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, or HIV or hepatitis B antigen
* Indicators of abnormal renal function at baseline: any urine protein
* History of allergy to Gamma-Secretase Inhibitor or related compounds
* History of any significant drug allergy
* Prior exposure to BMS-708163
* Exposure to any investigational drug or placebo within 4 weeks of study drug administration
* Use of any prescription drugs or over-the-counter acid controllers within 4 weeks prior to study drug administration
* Use of any other drugs, including over-the-counter medications and herbal preparations, within 2 weeks prior to study drug administration
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Within 30 days after the follow-up evaluation on Day 28

SECONDARY OUTCOMES:
Plasma concentration | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Yokohama, Kanagawa, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx